CLINICAL TRIAL: NCT03581799
Title: Investigation of Palatability of an Oral Dispersible Tablet (ODT) Formulation in Children Aged 2 to 10 Years
Brief Title: Palatability of an Oral Dispersible Tablet (ODT) Formulation in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-01367
Record Dates: First submitted 2018-06-21; First posted 2018-07-10 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Healthy
Keywords: Child

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral dispersible tablet (Other): 5 mm calcium carbonate based ODT will be administered by placing it in the buccal pouch (children aged 2-5 years) or on the tongue (children aged 6-10 years).
  Interventions: Other: Oral dispersible tablet

INTERVENTIONS:
Other: Oral dispersible tablet — Administration of a 5 mm calcium carbonate based ODT placed in the buccal pouch (children aged 2-5 years) or on the tongue (children aged 6-10 years).
  Other Names: Oral dispersible tablet (carrier tablet - no active pharmacological ingredient)

SUMMARY:
This is a cross-sectional study investigating the palatability of an oral dispersible tablet with no pharmacologically active agent (carrier tablet) in children without underlying acute or chronic disease aged 2 to 10 years of age.

DETAILED DESCRIPTION:
Oral dispersible tablets (ODTs) are a monolithic solid formulation potentially appropriate for a wide range of paediatric age groups. They also have a number of advantages over more frequently used formulation types, such as suspensions. Currently few Commercial products are available as ODTs for administration to children. Investigators aimed to investigate the palatability of an oral dispersible tablet with no pharmacologically active agent (carrier tablet) by assessing overall parent-reported, observer-reported and, where appropriate, child-reported acceptance of the formulation. In addition, investigators assessed the in situ disintegration behaviour of the carrier tablet.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 and 10 years
* Attending study site as an outpatient during the study period.
* Informed consent form for study participation signed by legal guardian
* Verbal assent to participation from child

Exclusion Criteria:

* Wearing dental braces
* Injuries or inflammatory disease affecting the oral cavity or throat
* Dysphagia
* Olfactory impairment
* Known renal impairment
* Known hypercalcaemia,
* Any known allergy against medications
* Ongoing antibiotic treatment at the time of the study
* Moderate-severe developmental delay as reported by the parents
* Parents/legal guardians are unlikely to reliably complete structured questionnaire because of significant language barriers
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Parent-reported palatability assessed by interview | Day 1
  5-point Likert scale, 1 "completely acceptable" to 5 "completely unacceptable"
Child-reported palatability (children aged 6-10 years only) assessed by interview | Day 1
  6-point Facial Hedonic Scale (0 "no discomfort on taking tablet" to 10 "maximum discomfort on taking tablet"

SECONDARY OUTCOMES:
Observer-reported palatability assessed by questionnaire | Day 1
  4-point Likert scale (0 "child refuses to take tablet" to 4 "child proactively takes tablet")
In-situ disintegration behaviour of carrier tablet | Day 1
  Staff-observed disintegration of the tablet at 20, 40 and 60 seconds of placement

CONTACTS AND LOCATIONS:
Overall Officials: Julia Bielicki, MD, Principal Investigator — University of Basel Children's Hospital
Locations (1):
- UKBB, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No